CLINICAL TRIAL: NCT05324280
Title: Acupuncture in a Multidisciplinary Approach for Vulvodynia and Chronic Pelvic Pain
Acronym: AMALIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Amalia V2.4.
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Vulvodynia; Chronic Pelvic Pain
Keywords: acupuncture
MeSH Terms: conditions — Vulvodynia | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Randomised controlled clinical study with waiting list control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Group (Experimental): Acupuncture treatment will be performed according to a defined protocol, and includes body and ear acupuncture. The needles will be stimulated manually and will remain for 20 minutes.
  Body acupuncture needles (diameter 0.3mm, length 30 mm) will be placed on the following positions:
  On the lower abdomen and back within Th11 and L1
  * Kidney 13 and 14; alternately unilaterally
  * Ren2 and 3 (midline) On classical acupuncture points on the extremities and the head
  * Stomach 36, Spleen 6; bilaterally
  * Large intestine 4, Liver 3; Bladder 60 bilaterally
  * Du 20 (midline)
  Ear acupuncture:
  Ear acupuncture needles (diameter 0,2 mm, length 20mm) will be used:
  Veg. I (Sympathetic), lower pelvis, hypogastric plexus, Heart,Thalamus, genital system (combining Chinese and French ear acupuncture)
  For point detection an electric potentiometer will be used. Ear points are punctured according to their generally accepted positions.
  Interventions: Procedure: Acupuncture
- Waiting list Group (No Intervention): Participants allocated to the waiting list control group may continue previously initiated standard therapy, but must not initiate any new treatment. They will be asked not to undergo acupuncture treatment for any condition within the next 3 months. After this period they are offered 10 acupuncture treatments over a period of 3 months.

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture treatment will be performed according to a defined protocol, and includes body and ear acupuncture.
  Arms: Acupuncture Group

SUMMARY:
Background: Vulvodynia and chronic pelvic pain (CPP) are common and challenging gynecologic pain syndromes. A multidisciplinary approach is recommended.

Study aim: To study the effectiveness of acupuncture as part of a multimodal treatment for women with vulvodynia and CPP.

Design: Randomised controlled clinical study

Study Population: Recruitment from a University outpatient clinic Study groups: Participants will be randomised (1:1)

* Acupuncture group
* Waiting list control group

Sample size: 68 patients

Study outcome

* Subjective Pain Perception (VAS)
* Health-related quality of life (questionnaires)

ELIGIBILITY:
Inclusion Criteria:

* Women with vulvodynia and/or chronic pelvic pain of at least 6 months duration
* multidisciplinary treatment for at least 3 months

Exclusion Criteria:

* Pregnancy
* Current malignancy
* Major neurologic or psychiatric morbidity
* Study participation in Lydia trial (Lasertherapy for vulvodynia)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change of Subjective Pain Perception | evaluation at 3 and 6 months
  Numeric Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst pain)

SECONDARY OUTCOMES:
Change of Health-related quality of life - DSF | evaluation at 3 and 6 months
  Questionnaire,German Pain Assessment (Deutscher Schmerzfragebogen/DSF). The modules on pain assessment (e.g. pain characteristics, relieving and aggravating factors) and on demographic information will be used.
Change of Health-related quality of life - PHQ-D | evaluation at 3 and 6 months
  Questionnaire Patient Health Questionnaire (PHQ-D) 9 is a sensitive screening tool for detecting depressive symptoms in a general patient population
Change of Health-related quality of life - PSQ | evaluation at 3 and 6 months
  Questionnaire Pain sensitivity questionnaire (PSQ) is an instrument for the assessment of pain sensitivity based on pain intensity self ratings of daily life situations
Change of Health-related quality of life - EHP-30 | evaluation at 3 and 6 months
  Questionnaire Endometriosis Health Profile (EHP-30) contains a total of 30 items. The modular part consists of six scales (work, relationship with children, sexual intercourse, infertility, medical profession, and treatment) and contains a total of 23 items. Items within scales are summed to create a raw score, and then each scale is translated into a score ranging from 0 (best health status) to 100 (worst health status)
Change of Subjective improvement | evaluation at 3 and 6 months
  Patient Global Impression of Improvement (PGI-I) scale is a ), a single item instrument with a 7-step Likert type response scale to assess subjective improvement after treatment
Patient treatment satisfaction | evaluation at 3 months
  "Fragebogen zur Patientenzufriedenheit - ZUF8" is an 8-item tool for measuring global patient satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology/ Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No